CLINICAL TRIAL: NCT01824966
Title: Signet Ring Cells in Esophageal and GE Junction Carcinomas Have a More Aggressive Biological Behavior
Brief Title: Signet Ring Cell Carcinoma in Esophageal Adenocarcinoma
Acronym: SRCC
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, RN, MSc, Datamanager, University Hospital, Gasthuisberg
Other Study IDs: SRCC
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Adenocarcinoma; Esophageal Cancer
Keywords: Esophagectomy; Signet Ring Cells
MeSH Terms: conditions — Adenocarcinoma; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SRC<50%: Adenocarcinoma containing < 50% of signet ring cells
- SRC>50%: Adenocarcinoma containing > 50% of signet ring cells

SUMMARY:
There has been much controversy surrounding the biologic behavior and prognosis of esophageal signet ring cell (SRCs) containing carcinomas. To clarify the biologic behavior of SRCs, the investigators compared the clinicopathologic features and prognosis of SRCs with other adenocarcinomas (ADC) of the esophagus and gastroesophageal junction (GEJ).

DETAILED DESCRIPTION:
Adenocarcinoma (ADC) of the esophagus and gastroesophageal junction (GEJ) is an aggressive neoplasm and has a poor prognosis. Surgical based treatment has been the treatment of choice for localized esophageal adenocarcinoma.

Signet-ring cell carcinoma is a unique histologic subtype of adenocarcinoma characterized by abundant intracellular mucin accumulation and a compressed nucleus displaced toward one extremity of the cell (the so-called signet-ring cell (SRC)). According to the World Health Organisation (WHO), a true signet-ring cell carcinoma (SRCca) is defined as an adenocarcinoma in which the predominant component (more than 50% of the tumor) consists of isolated or small groups of SRC in the stroma. If the tumor contains less than 50% of those cells, it is generally considered as an adenocarcinoma (ADC).

ELIGIBILITY:
Inclusion Criteria:

- Adenocarcinoma R0 resection Primary surgery

Exclusion Criteria:

- Other histology R1 or R2 resection Neoadjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From our prospectively built database we retrieved all adenocarcinoma from 1990 till 2009 who underwent primary surgery with R0 resection. Seven hundred seventy-nine patients were included for further analysis. Pathology reports mentioning signet ring cells (n = 82) were reviewed by our pathologist and, after confirmation, tumors were classified into two groups according to WHO criteria (>50% SRC or <50% SRC). The remaining 697 ADC patients served as control group.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cancer specific 5 year survival in SRCC | from surgery
  Cancer specific 5 year survival classified into two groups according to WHO criteria (>50% SRC or <50% SRC)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nafteux, MD, Principal Investigator — University Hospital Leuven; Dept. of Thoracic Surgery
Locations (1):
- University Hospital Leuven; Dept. of Thoracic Surgery, Leuven, Belgium